CLINICAL TRIAL: NCT01603771
Title: Neural Activation and Connectivity in Response to Exercise and Cognitive Training
Acronym: NAC
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201104290; 7432-01 (Other Grant/Funding Number: Barnes Jewish Hospital Foundation)
Record Dates: First submitted 2012-05-02; First posted 2012-05-23 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Neural Connectivity
Keywords: Adult; Exercise; Cognition; MRI
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Combined: Participants assigned to this group have been randomized to the Combined group of the parent study, Combining Exercise and Cognitive Training to Improve Everyday Function(EXACT)(Unique Protocol ID 201102416). Participants perform a 6-month standardized aerobic training program at a local recreational center, 3 times per week for 1 hour. Participants in this group also perform an 8-week cognitive training program 3 days per week for 1 hour, during months 5 and 6. The cognitive training program is computer-based, and focuses on 3 types of cognitive processes: task coordination, prospective memory, and retrospective memory retrieval. The cognitive training is conducted on concurrent days with aerobic exercise training sessions, also on site at the recreational center.
  Interventions: Other: Blood Oxygen Level Dependent (BOLD) functional magnetic imaging (fMRI)
- Control: Participants assigned to this group have been randomized to the Control group of the parent study, Combining Exercise and Cognitive Training to Improve Everyday Function(EXACT)(Unique Protocol ID 201102416). Participants perform a 6-month home exercise program consisting of stretching, range of motion, and simple yoga exercises designed to improve flexibility. They are instructed to perform these exercises at home at least 3 times per week for 30 - 45 minutes and record their activity on a calendar. Participants also attend weekly 1-hour Health Education sessions for 8 weeks, during months 5 and 6. These sessions cover topics unrelated to exercise or cognition, such as nutrition, hearing loss, stroke, and home energy conservation.
  Interventions: Other: Blood Oxygen Level Dependent (BOLD) functional magnetic imaging (fMRI)

INTERVENTIONS:
Other: Blood Oxygen Level Dependent (BOLD) functional magnetic imaging (fMRI) — All participants complete MRI scans at baseline and at the end of month 6. Scanning sessions last approximately 30 minutes each and consist of two components: (1) High resolution T1-weighted MPRAGE anatomic images to provide detailed anatomy and maximum gray-white matter contrast for images and to allow any estimate of regional or whole-brain volume, and (2) Resting BOLD functional images to allow assessment of the functional connectivity in large scale networks.

SUMMARY:
The goal of this pilot study is to evaluate whether healthy, sedentary older adults have increased activation of specific brain areas, in response to exercise and cognitive training, in comparison to a control group, and whether improvements in psychometric test performance are related to increased activation of brain networks. Participants, between age 55-75 years will be recruited from an ongoing study of exercise and cognitive training, to undergo Blood Oxygen Level Dependent (BOLD) functional magnetic imaging (fcMRI).

ELIGIBILITY:
Inclusion Criteria:

* meet the inclusion criteria for the parent study, Combining Exercise and Cognitive Training to Improve Everyday Function (EXACT) study (Unique Protocol ID 201102416).

Exclusion Criteria:

* currently taking chronic psychotropic medication, beta blockers, or calcium channel blockers
* contraindication to MRI scanning
* inability to complete MRI scans in closed scanner

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will include 24 adults, male and female, aged 55-75 years who meet eligibility criteria for and are enrolled in the parent study, Combining Exercise and Cognitive Training to Improve Everyday Function (EXACT), Unique Protocol ID 201102416. Participants will be sedentary (not exercising regularly) but otherwise generally healthy.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Functional connectivity of large-scale brain networks as seen through Blood Oxygen Level Dependent (BOLD) functional magnetic resonance imaging (fMRI) | Change in connectivity measurements between baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ellen F. Binder, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States